CLINICAL TRIAL: NCT05190406
Title: Success and Quality of Life Following Complete Pulpotomy and Root Canal Treatment in Teeth With Clinical Signs Indicative of Irreversible Pulpitis
Brief Title: Success and Quality of Life Following Complete Pulpotomy and Root Canal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kanagadurga
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Irreversible Pulpitis
Keywords: pulpitis; pulpotomy; single visit root canal treatment; bioceramic material
MeSH Terms: conditions — Pulpitis | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): complete pulpotomy will be done till the level of root canal orifice.
  Interventions: Procedure: Pulpotomy
- Root canal treatment (Active Comparator): Single visit root canal treatment will be done according to standard protocol.
  Interventions: Procedure: root canal treatment

INTERVENTIONS:
Procedure: Pulpotomy — After achieving hemostasis, in pulpotomy group bioceramic material will be placed and then permanent restoration will be done.
  Arms: Pulpotomy
Procedure: root canal treatment — Single visit root canal treatment will be done according to standard protocol.
  Arms: Root canal treatment

SUMMARY:
The purpose of this study is to compare the Success and quality of life following complete pulpotomy and root canal treatment in teeth with clinical signs indicative of irreversible pulpitis.

DETAILED DESCRIPTION:
After thorough history and clinical and radiographic examination, and confirmation of eligibility for the study, risks and benefits associated with the procedure will be explained and written informed consent will be taken from the patients. Study subjects will be randomly allocated to either Complete pulpotomy or Root canal treatment Group.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent restorable mandibular molar teeth.
* Tooth should give positive response to pulp sensibility testing.
* Clinical diagnosis of irreversible pulpitis with PAI score≤2.
* Tooth with probing pocket depth and mobility are within normal limits.
* Non-contributory medical history.

Exclusion Criteria:

* Teeth with immature roots.
* No pulp exposure after caries excavation.
* Bleeding could not be controlled in 6 minutes.
* Insufficient bleeding after pulp exposure, the pulp is judged necrotic or partially necrotic.
* Absence of antagonist tooth.
* Positive history of antibiotic use in the past 1 month or requiring antibiotic prophylaxis
* Had taken analgesic in past 3 days.
* Tooth with periapical lesion visible on radiograph

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | 6 months and one year
  Clinical success criteria No history of spontaneous pain No tenderness to palpation or percussion Normal mobility and probing pocket depth. Soft tissues around tooth are normal with no swelling or sinus tract.
Radiographic success rate | 6 months and one year
  Radiographic success criteria No pathosis evident on the radiograph Periapical Index score 1 or 2

SECONDARY OUTCOMES:
Oral Health related quality of Life | baseline to one week, 6 months and one year
  Oral Health Impact Profile-14 questionnaire of score 0-4 will be used to assess the quality of life. Score 0 means never and 4 means very often affected the quality of life.
Pain assessment | baseline to one week
  Visual analogue Scale of 0 to 10 Centimetere line will be used to assess pain. Score 0 means no pain and Score 10 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Tewari, MDS, Study Director — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK, Haryana, India, 124001
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India